CLINICAL TRIAL: NCT02917343
Title: Effect of Mirror Therapy and Repetitive Task Training on Upper Extremity Function for Persons With Subacute Stroke
Brief Title: Effect of Mirror Therapy and Task Oriented Training for Persons With Paretic Upper Extremity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quinnipiac University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2614
Record Dates: First submitted 2016-09-26; First posted 2016-09-28 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Stroke; Cerebrovascular Accident
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intervention arm (Experimental): participants received 4 weeks of mirror therapy and repetitive task training
  Interventions: Behavioral: mirror therapy and repetitive task training

INTERVENTIONS:
Behavioral: mirror therapy and repetitive task training
  Other Names: task oriented training

SUMMARY:
The purpose of the study is to determine the effect of a combined mirror therapy and task oriented/repetitive task training on upper extremity function of persons with hemiplegia due to cerebrovascular accident or stroke.

DETAILED DESCRIPTION:
This case series was designed to to determine the effect of a mirror therapy and repetitive task training program on the weak arm and hand functioning due to the consequences of stroke. Mirror therapy is a type of therapy mirror reflection of the stronger arm and hand helps to promote reorganization of neurons. Studies have shown that mirror therapy is an effective adjunct to regular exercise and task-oriented therapy.

To qualify for this study, participants must meet the following criteria: 1) age 21 years or more; 2) first-time stroke with onset of at least 3 months; 3) slight movement of the weaker arm or /and hand; 3) stable physical and mental health; and 4) mentally capable and competent to make health care-related decisions and carry out a home program.

Participants were required to come to Quinnipiac University - North Haven campus to undergo mirror therapy training, in 45-60 minute sessions, twice a week for one month. They were also required to complete pre-testing before and post-testing after the mirror therapy program. In addition, they were required to carry-out a home program that includes the use of a mirror box and self-selected tasks. The home program required them to exercise and practice the use of their more affected arm and hand for at least 1-2 hours a day.

Participation was strictly voluntary. Participants were informed of the minimal risks involved as well as their options to continue or withdraw from the study upon initial consent. The study did not yield physical or mental harm to the participants.

ELIGIBILITY:
Inclusion Criteria:

* able to give consent, complete home program
* minimal arm and hand use with the paretic limb
* onset of stroke of at least 3 months

Exclusion Criteria:

* >1 stroke episode
* significant cognitive and visual perceptual deficit
* lack of social support

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in Patient Specific Functional Scale | Change from baseline at 2 months
  Patient Specific Functional Scale is a measure that involves self-rating of self-selected functional tasks
Change in Fugl Myer Motor Assessment | Change from baseline at 2 months
  Fugl-Meyer Motor Assessment is a clinical performance test of motor ability of the upper extremity

SECONDARY OUTCOMES:
Change in Motor Activity Log | Change from baseline at 2 months
  The Motor Activity Log is a self-reported measure that captures the amount of arm and hand use and perception of movement quality of the impaired upper limb

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Bondoc S, Booth J, Budde G, Caruso K, DeSousa M, Earl B, Hammerton K, Humphreys J. Mirror Therapy and Task-Oriented Training for People With a Paretic Upper Extremity. Am J Occup Ther. 2018 Mar/Apr;72(2):7202205080p1-7202205080p8. doi: 10.5014/ajot.2018.025064. PMID 29426386